CLINICAL TRIAL: NCT03358550
Title: Influence of an Imaginary Target on the State of Accommodation Under Scotopic Conditions
Brief Title: Night Myopia and Dark Focus of Accommodation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences Jena (Other)
Responsible Party: Principal Investigator, Philipp Hessler, Principal Investigator, University of Applied Sciences Jena
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UASJena
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Dark Focus of Accommodation
Keywords: accommodation; dark focus; night myopia

STUDY DESIGN:
Masking Description: Sequence of tests was randomized. It is no multi-arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accommodation in scotopic luminance (Experimental)
  Interventions: Diagnostic Test: Accommodation Measurement

INTERVENTIONS:
Diagnostic Test: Accommodation Measurement — Accommodation was measured for different distances and light conditions.

SUMMARY:
Shifts in accommodation at decreasing luminance levels are considered as principle cause for night myopia. Previous studies with laser optometers quantified the dark focus of accommodation up to 3 D. In addition to the measurement of dark focus, the aim of this study was to investigate the influence of an imaginary target at finite distances on the state of accommodation at scotopic luminance.

DETAILED DESCRIPTION:
Accommodation was measured by using an open-field autorefractor (WAM 5500, GRAND SEIKO). Full corrected right eyes of 39 subjects aged from 18 to 40 years were investigated in this randomized, cross-sectional study. Accommodation measurements in photopic luminance were taken for 6 m of empty field and for optotype fixation at 2 m, 1 m and 0.5 m. At scotopic luminance, dark focus of accommodation was examined directly after darkening and after 10 min of dark adaptation. After adaptation, subjects had to visualize imaginary targets in the four distances while accommodation was measured.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 44
* visual acuity at least 0.8 (5/6)

Exclusion Criteria:

* medication with an impact on the visual system
* visual disease or disease with an impact on the visual system
* pregnancy or other hormonal variances
* drug usage
* overfatigue at the period of investigation
* mental handicap

Ages: 22 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Shift of accommodation in scotopic luminance (Dark focus) | Baseline only
  Accommodative shift in scotopic luminance compared to photopic luminance for empty field (dark focus of accommodation)

SECONDARY OUTCOMES:
Difference of accommodation for 2 m target | Baseline only
  Accommodative shift in scotopic luminance compared to photopic luminance for the fixation of a target in 2 m
Difference of accommodation for 1 m target | Baseline only
  Accommodative shift in scotopic luminance compared to photopic luminance for the fixation of a target in 1 m
Difference of accommodation for 0.5 m target | Baseline only
  Accommodative shift in scotopic luminance compared to photopic luminance for the fixation of a target in 0.5 m

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Hessler, M.Sc., Principal Investigator — University of Applied Sciences Jena
Locations (1):
- University of Applied Sciences, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No